CLINICAL TRIAL: NCT06914388
Title: Effects of Self-Management Strategies on Pain, Muscle Stiffness and Temporomandibular Joint Functions in Individuals With Bruxism
Brief Title: Impact of Self-Management Strategies in Self-Reported Bruxism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cyprus International University (Other)
Responsible Party: Principal Investigator, Mehmet Miçooğulları, Asst. Prof. Dr., Cyprus International University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 020-5790
Record Dates: First submitted 2025-03-28; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Bruxism; Self-management; Pain; Proprioception; Temporomandibular Joint Dysfunction
Keywords: Bruxism; Self-Management Strategies; Proprioception; Muscle Stiffness; Pain; Temporomandibular Joint Dysfunction
MeSH Terms: conditions — Bruxism; Pain; Temporomandibular Joint Disorders

STUDY DESIGN:
Intervention Model Description: Interventional Study
Masking Description: All treatments were administered by the same physiotherapist. All assessments were carried out by a physiotherapist who was blinded to the treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Self-Management (Experimental): Participants were recruited from individuals seeking treatment at a physiotherapy clinic.
  Interventions: Other: Self-Management Strategies

INTERVENTIONS:
Other: Self-Management Strategies — Stretching exercises, strengthening exercises, massage, relaxing exercises, breathing exercises, patient education

SUMMARY:
This study aim to evaluate the effects of a 6-week self-management program on pain, muscle stiffness, and temporomandibular joint (TMJ) functions in sedentary individuals aged 18-40 with bruxism. Thirty-five individuals will be evaluated. Bruxism will be assessed using the Bruxism Assessment Questionnaire, while temporomandibular joint dysfunction (TMJD) will be evaluated using the Helkimo Clinical Dysfunction Index and the Fonseca Questionnaire. Masseter muscle pain threshold will be measured with a digital algometer, muscle stiffness with a Shore Durometer, mandibular depression range of motion with a bicondylar caliper, and TMJ proprioception with TMJ position sense. Assessments will be conducted pre-intervention and at the end of the fourth week.

DETAILED DESCRIPTION:
The 4-week self-management program significantly increased the masseter pain threshold (p<0.001) and reduced muscle stiffness at rest and during contraction (p<0.001). TMJD severity, as measured by the Helkimo Index (p=0.010) and Fonseca Questionnaire (p<0.001), was significantly reduced. Additionally, TMJ position sense and mandibular depression range of motion improved significantly (p<0.001). Self-management strategies positively impact bruxism symptoms, including pain, muscle stiffness, and TMJ functions. These strategies should be considered an integral part of TMJD and bruxism management.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 40 years
* Sedentary lifestyle
* Clinical diagnosis of sleep and/or awake bruxism

Exclusion Criteria:

* Significant musculoskeletal disorders of the cervical or thoracic spine
* Chronic illnesses
* Neurological conditions affecting balance and postural control
* Pregnancy
* The presence of dental prostheses
* Participants who missed more than 15 sessions

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2024-07-03 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2025-02-17 (Actual)

PRIMARY OUTCOMES:
Bruxism Assessment | 8 weeks
  Bruxism will be assessed using self-reports, which are considered appropriate for both clinical and research purposes. Awake bruxism will be diagnosed based on participants' self-awareness, determined by asking whether they had noticed clenching or grinding their teeth while awake in the past six months. Individuals who respond affirmatively will be classified as having awake bruxism. Sleep bruxism will be diagnosed using the 2014 criteria established by the American Academy of Sleep Medicine (AASM). Participants will be asked whether they frequently noticed teeth grinding during sleep, will be informed of it by others, or observed excessive tooth wear. Additionally, they will be questioned about symptoms upon waking, such as jaw fatigue, tension, or pain; sensations of clenching or pain in the mouth; temple pain; difficulty opening the mouth; tension in the jaw joint requiring movement to release; or clicking sounds in the jaw joint that disappear afterward.
Temporomandibular Joint Dysfunction | 8 weeks
  Temporomandibular Joint Disorder (TMJD) will be evaluated using the Helkimo Clinical Dysfunction Index (HCDI). This instrument is considered valid and reliable measures of TMJD. The scoring system categorises participants into four groups: no clinical symptoms (score 0), mild TMJD (scores 1-4), moderate TMJD (scores 5-9), and severe TMJD (scores 10-25)
Temporomandibular Joint Dysfunction | 8 weeks
  Temporomandibular Joint Disorder (TMJD) will be evaluated using the Fonseca Questionnaire. This instrument is considered valid and reliable measures of TMJD. Participants will be instructed to respond to each question as 'yes' (10 points), 'no' (0 points), or 'sometimes' (5 points). The questionnaire results will be classified as no TMJD (0-15), mild TMJD (20-40), moderate TMJD (45-65), and severe TMJD (70-100) based on the responses provided by the participants.
Masseter Muscle Pain Threshold Measurement | 8 weeks
  The pain threshold of the masseter muscle will be assessed bilaterally over the muscle belly using a JTECH Commander digital algometer. Three measurements will be taken from the muscle belly, and the average value will be calculated. Participants will be instructed to indicate the moment they first perceived pain, and the value will be display on the device will be recorded as the pain threshold in pounds. Higher scores indicate better pain threshold.
Masseter Muscle Stiffness | 8 weeks
  The stiffness of the masseter muscle will be assessed using a Shore Durometer OO (M&A Instruments Inc., United States), a handheld device designed for convenient and non-invasive measurement of muscle stiffness. The durometer evaluates tissue properties by measuring oscillations generated through mechanical contact with the assessed muscle. Measurements will be performed bilaterally over the belly of the masseter muscle during both resting and maximum contraction states. Each measurement will be repeated three times, and the average values will be recorded in Newtons per meter.

SECONDARY OUTCOMES:
Temporomandibular Joint Position Sense | 8 weeks
  The measurement of TMJPS will be conducted using 9 test sticks ranging from 4 mm to 8 mm in thickness, with 0.5 mm increments. A 6 mm thick wooden bar will be used as a reference. Participants first bit the 6 mm reference stick with their front teeth for 1 minute to familiarize themselves with the reference thickness. Subsequently, they will be asked to bite each of the 9 test sticks in a random order and compare their thickness to the reference stick. Each test stick will be presented 5 times, resulting in a total of 45 tests. Participants will indicate whether the test stick felt "thinner," "thicker," or "equal" compared to the reference stick. During the test, participants' eyes will be closed, and their responses will be recorded as correct (1 point) or incorrect (0 points). Total scores will be calculated for analysis.
Mandibular Depression Range of Motion | 8 weeks
  The range of motion for mandibular depression will be assessed by evaluating the maximum mouth opening. Participants will be instructed to open their mouths as wide as possible. The distance between the lower and upper central incisors will be measured using a bicondylar caliper (Holtain Ltd., UK) and will be recorded in centimeters (cm). Each measurement will be repeated three times, and the average value will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Salih Angın, Prof. Dr., Study Chair — Cyprus International University
Locations (1):
- Turkey, Mersin, Lefkosa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mesko ME, Hutton B, Skupien JA, Sarkis-Onofre R, Moher D, Pereira-Cenci T. Therapies for bruxism: a systematic review and network meta-analysis (protocol). Syst Rev. 2017 Jan 13;6(1):4. doi: 10.1186/s13643-016-0397-z. PMID 28086992
- [Background] Micoogullari M, Yuksel I, Angin S. Efficacy of scapulothoracic exercises on proprioception and postural stability in cranio-cervico-mandibular malalignment: A randomized, double-blind, controlled trial. J Back Musculoskelet Rehabil. 2024;37(4):883-896. doi: 10.3233/BMR-230323. PMID 38427467
- [Background] Winocur E, Uziel N, Lisha T, Goldsmith C, Eli I. Self-reported bruxism - associations with perceived stress, motivation for control, dental anxiety and gagging. J Oral Rehabil. 2011 Jan;38(1):3-11. doi: 10.1111/j.1365-2842.2010.02118.x. PMID 20557433
- [Background] Koyano K, Tsukiyama Y, Ichiki R, Kuwata T. Assessment of bruxism in the clinic. J Oral Rehabil. 2008 Jul;35(7):495-508. doi: 10.1111/j.1365-2842.2008.01880.x. PMID 18557916
- [Background] Manfredini D, Bucci MB, Sabattini VB, Lobbezoo F. Bruxism: overview of current knowledge and suggestions for dental implants planning. Cranio. 2011 Oct;29(4):304-12. doi: 10.1179/crn.2011.045. PMID 22128671
- [Background] Feu D, Catharino F, Quintao CC, Almeida MA. A systematic review of etiological and risk factors associated with bruxism. J Orthod. 2013 Jun;40(2):163-71. doi: 10.1179/1465313312Y.0000000021. PMID 23794697